CLINICAL TRIAL: NCT07207057
Title: Edmond J Safra, Accelerating Clinical Trials in Parkinson's Disease (EJS ACT-PD) - a Multi-arm Multi-stage Platform Trial for Potential Disease Modifying Approaches.
Brief Title: Edmond J. Safra Accelerating Clinical Trials in Parkinson's Disease: A Multiarm Multi-stage Platform Trial
Acronym: EJS ACT-PD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cure Parkinson's (Other); Parkinson's UK (Other); National Institute for Health Research, United Kingdom (Other Government); John Black Charitable Foundation (Unknown); Medical Research Council (Other Government); Newcastle University (Other); Van Andel Research Institute (Other); Michael J. Fox Foundation for Parkinson's Research (Other); Gatsby Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND002; ISRCTN17799294 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2025-05-09; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Parkinsons Disease (PD)
MeSH Terms: conditions — Parkinson Disease | interventions — Telmisartan; Terazosin

STUDY DESIGN:
Intervention Model Description: Multi-arm multi-stage (MAMS) trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As the trial is double-blinded, neither participants nor delivery staff will be aware of which treatment a participant has been randomised to. Participants' treatment allocations will be stored only in the randomisation server, separate to the EJS ACT-PD Trial database There will be a Trial Statistician at the MRC CTU at UCL who will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Arm A) (Placebo Comparator): Standard of Care (SoC) plus placebo.
  Interventions: Drug: Placebo
- Telmisartan (Arm B) (Experimental): Standard of Care (SoC) plus telmisartan
  Interventions: Drug: Telmisartan
- Terazosin (Arm C) (Experimental): Standard of Care (SoC) plus terazosin
  Interventions: Drug: Terazosin (Hytrin)

INTERVENTIONS:
Drug: Placebo — An over-encapsulated placebo capsule taken once daily to match the treatment arms following a 5-week titration phase.
  Arms: Placebo (Arm A)
Drug: Telmisartan — Over-encapsulated telmisartan 40mg per day for 36 months (plus their usual SoC) following a 5-week titration phase.
  Titration phase for telmisartan: Week 1-3: one 20 mg capsule per day; Week 4-5: one 40 mg capsule per day
  Arms: Telmisartan (Arm B)
Drug: Terazosin (Hytrin) — Over-encapsulated terazosin 5mg per day for 36 months (plus their usual SoC) following a 5-week titration phase.
  Titration phase for terazosin: Week 1: one 1 mg capsule per day; Week 2: one 2 mg capsule per day; Week 3: one 3 mg capsule per day; Week 4: one 4 mg capsule per day; Week 5: one 5 mg capsule per day
  Arms: Terazosin (Arm C)

SUMMARY:
Parkinson's disease (PD) is currently the fastest-growing neurological condition globally. It is projected to affect 172,000 people in the UK by 2030,with the current annual cost to the country being ~£3.6 billion. The disease progressively impairs physical abilities, leading to increased disability, falls, and difficulties with speech, swallowing, mood, thinking, and memory. While existing treatments can alleviate some symptoms, their effectiveness diminishes over time, and they can cause severe side effects. This trial uses a Multi-Arm,Multi-Stage (MAMS) design where multiple treatments are tested simultaneously in separate groups, called "arms." Each treatment is compared against a placebo, a dummy treatment with no active ingredients, to evaluate its effectiveness and safety. Throughout the trial, each treatment undergoes periodic reviews, known as interim analyses, to assess its safety and potential benefits. If a treatment shows promise, it continues in the trial until a final assessment determines its overall effectiveness. Treatments that do not show positive results are discontinued and replaced with new candidates. This approach reduces the number of participants needed to obtain reliable results and is more cost-effective and faster than conducting separate trials for each treatment. The treatments selected for this trial were chosen based on careful consideration of existing evidence regarding their safety and effectiveness. To choose the treatments we want to test, we carefully considered evidence for safety and effectiveness. The trial will start with two treatment arms (telmisartan and terazosin) and one placebo arm, with a third treatment arm added after one year. We can identify new treatments to add to the trial each year. Participants will be followed up for up to 36 months. After an in-person screening visit, all remaining visits at 3 months,6 months and then every 6 months after, for a total of up to 36 months can be completed remotely. The visits will include questionnaires, assessment of Parkinson's symptoms and discussions about any side effects. Participants will informed of trial progress. Results will be shared via the trial website and published in a medical journal.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis by neurologist, movement disorders specialist or appropriately experienced clinician of clinically established or clinically probable PD in the clinician's opinion. In the presence of any diagnostic doubt, the Movement Disorder Society diagnostic criteria will be applied.
2. Diagnosed with Parkinson's disease at age 30 years or older, no upper age limit.
3. Currently on Parkinson's medication (levodopa-containing preparations or dopamine agonists, used either as single agents or in combination) for at least 2 months prior to screening visit.
4. Female participants who are women of child-bearing potential (WOCP) must have confirmation of a negative pregnancy test at screening visit.
5. Female participants who are WOCP and male participants and their partners who are WOCP must be taking highly effective contraceptive treatment(s).
6. Documented informed consent.
7. Eligible for at least one of the active treatment arms (See treatment specific exclusions).
8. Randomisation should ideally take place within 3 weeks of the screening visit but no later than 4 weeks after the screening visit.
9. If a participant is being re-randomised into the trial, additional timing of entry requirements must also be met:

   * For participants being re-randomised after completing 36 months' follow-up and the arm was not closed due to lack of activity, a 26-week washout period from last dose of IMP must be completed before their screening visit. If the primary analysis indicates that the IMP was ineffective then this washout period can be reduced to 6 weeks.
   * For participants being re-randomised following treatment arm termination due to lack of activity, a 6-week washout period from their last dose of IMP must be completed prior to screening assessment.

Exclusion Criteria:

1. Diagnosis or suspicion of other cause for parkinsonism such as atypical parkinsonism, dystonic tremor, essential tremor, drug-induced parkinsonism.
2. Known carriers of recessive PD gene mutations PRKN, PINK1 or DJ1 (based on previous medical tests / notes).
3. Clinical diagnosis of dementia or MoCA <21 at screening visit.
4. Currently in another ongoing interventional trial or exposure to any IMP within an experimental interventional trial within 6 months prior to screening visit (exception for EJS ACT-PD participants that are being re-randomised due to treatment arm termination following lack of activity as only a 6-week wash out period is required).
5. Unable or unwilling to comply with study requirements.
6. Diagnosis of clinically significant depression or >14 on PHQ-9 at screening visit.
7. Current suicidal ideation within one year prior to the screening visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS).
8. Previous brain surgery or on a waiting list for brain surgery including deep brain stimulation and / or currently taking or on a waiting list for advanced therapies for Parkinson's disease (such as any infusion therapy).
9. Monotherapy with monoamine oxidase-B inhibitor (MAO-BI).
10. Previous exposure to any of the currently recruiting IMPs within 6 months prior to screening visit or previous intolerance of any of the IMPs.
11. Participant has any concurrent medical condition, abnormal laboratory tests, progressive neurological disorder or uncontrolled, clinically significant systemic disease that, in the opinion of the Investigator, could cause study participation to be detrimental to the participant (e.g., end stage renal failure, severe heart failure, unstable angina, uncontrolled hypertension or uncontrolled orthostatic hypotension, severe liver disease, uncontrolled diabetes, or severe anaemia).
12. Pregnant or breastfeeding or intending to become pregnant during the study or within 70 days after the final dose of study drug.
13. Confirmed diagnosis of cancer and is requiring active management of that cancer and/or in the view of the local team, the diagnosis and/ or its treatment may compromise their ability to remain participating in the trial for 36 months or tolerate any of the active treatments.
14. Participants with hepatobiliary disorders or abnormal liver function tests at the screening visit consisting of one of the following:

    * ALT or AST >2x the upper limit of normal
    * Total serum bilirubin >1.5x ULN (except for participants with Gilbert's disease, for whom the upper limit of serum bilirubin is 51.3 μmol/l or 3mg/dl)
15. Participants with a history of alcohol/drug abuse/dependence within the 3 years prior to screening visit.
16. Participants with either of the following:

    * Sitting systolic blood pressure (SBP) less than 100 mmHg or sitting diastolic blood pressure (DBP) less than 50 mmHg, irrespective of symptoms
    * Orthostatic hypotension defined as any of the following:

      * Decrease in BP > 20 mmHg systolic or > 10 mmHg diastolic on supine to standing, associated with clinical symptoms
      * Decrease in BP >30mmHg systolic and/or BP >15 mmHg diastolic on supine to standing regardless of symptoms
      * If the lowest BP on standing is less than 100 mmHg or lowest diastolic on standing is less than 50 mmHg If, in the assessing clinician's opinion, the postural BP drop is attributable to transient/reversible factors (e.g. related to use of antihypertensives, dehydration, elevated room temperature, postprandial state), one repeated orthostatic BP assessment is allowed once those factors are addressed; additional re-screening will be allowed if the participant has their hypotension/orthostatic hypotension treated.

TREATMENT-SPECIFIC EXCLUSION CRITERIA

In addition to the core inclusion and exclusion criteria above, there are arm-specific eligibility criteria for each arm to determine to which arms a participant can be randomised:

Telmisartan-specific exclusion criteria

1. Participants currently taking sartans (AT1 angiotensin receptor antagonists), aliskiren, ACE inhibitors or potassium sparing diuretics.
2. Participants with a known hypersensitivity or intolerance to sartans (AT1RAs)
3. Participants with a history of angioedema.
4. Participants with known aortic or mitral stenosis that the investigator judges to make telmisartan use potentially unsafe.
5. Participants with known renal artery stenosis.
6. Participants with hyperkalaemia (serum potassium (K+) level of ≥ 5.5 mmol/l). If hyperkalaemia is identified, one re-screening will be allowed, either within 4 weeks or after identification and treatment of precipitants.
7. Participants currently taking lithium or taken within the previous 6 months.

Terazosin-specific exclusion criteria

1. Participants currently using alpha blockers other than tamsulosin (alfuzosin, silodosin, prazosin, terazosin, and doxazosin), including natural supplements with this action (e.g. yohimbine).
2. Participants with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
3. Participants with a known sensitivity to quinazolines e.g. alfuzosin, silodosin, prazosin, terazosin, and doxazosin, erlotinib, gefitinib, afatinib, lapatinib, and vandetanib.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I and II combined | baseline, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination and week 165
  The rate of Parkinson's disease progression between the active treatment and placebo arms is measured by the MDS-UPDRS Parts I and II combined with equal weighting

SECONDARY OUTCOMES:
Hoehn and Yahr Scale (H&Y) | screening, week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination and week 165
  Clinician reported measures. Parkinson's disease stage is measured using the Hoehn and Yahr Scale (H&Y)
Montreal Cognitive Assessment (MoCA) | screening, week 0, week 26, week 52, week 104, week 156 or early termination.
  Clinician reported measures. Cognitive impairment is measured using the Montreal Cognitive Assessment (MoCA)
levodopa-equivalent daily dose (LEDD) | all study visits
  Clinician reported measures. Parkinson's disease medication use is measured by levodopa-equivalent daily dose (LEDD).
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Remote) | screening, week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination and week 165.
  Clinician reported measures. Part III of the MDS-UPDRS in the ON medication state (remote elements only)
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV | screening, week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination and week 165
  Clinician reported measures. Part IV of the MDS-UPDRS in the ON medication state
Severity of depression | screening, week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. The severity of depression is assessed by the Patient Health Questionnaire (PHQ-9)
Quality of Life - Parkinson's Disease Questionnaire (PDQ-8) | week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. Quality of life is assessed by the Parkinson's Disease Questionnaire (PDQ-8)
Carers' quality-of-life assessed by the questionnaire for parkinsonism (PQoL Carers) | week 0, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. Carers' quality-of-life is assessed by the questionnaire for parkinsonism (PQoL Carers)
Ability to enjoy life (ICECAP-O) | week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. Ability to enjoy life is assessed by the ICEpop CAPability measure for Older people (ICECAP-O)
Health-related quality of life (EQ-5D-5L) | week 0, week 13, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. Health-related quality of life is assessed by the EuroQol five-dimension scale questionnaire (EQ-5D-5L). Has 5 response levels (no problems, some problems, moderate problems, severe problems, extreme problems) and a visual analogue scale capturing overall health (100 means the best health you imagine; 0 means the worst health you can imagine).
Use of health and social care resources | week 0, week 26, week 52, week 78, week 104, week 130 and week 156.
  Participant reported measures. Use of health and social care resources is assessed by the resource use questionnaire to determine participants use of different health services and the care and support received.
Carer health-related quality of life (EQ-5D-5L) | week 0, week 26, week 52, week 78, week 104, week 130, week 156 (end of study visit) or early termination.
  Participant reported measures. Carer health-related quality of life is assessed by the EuroQol five-dimension scale questionnaire (EQ-5D-5L)
Suicidal ideation (C-SSRS) | screening, week 156 (end of study visit) or early termination
  Safety and tolerability. Suicidal ideation is assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Adverse Events (Safety and Tolerability) | week 0, week 1, week, 2, week, 3, week 4, week 5, week 13, week 26, week 39, week 52, week 65, week 78, week 104, week 130, week 156, week 165
  Safety and tolerability. Other safety and tolerability measures are assessed through the collection of adverse events/serious adverse events, treatment compliance and trial withdrawal and treatment discontinuation rates
Participant experience of trial participation | week 0, week 78, week 156 (end of study) or early termination
  Participant experience before, during and after trial participation as assessed by the Study Participant Feedback Questionnaire (SPFQ), which includes written feedback and responding to statements using the responses: Strongly disagree, Disagree, Neither agree or disagree, Agree and Strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Thomas Foltynie, Principal Investigator — University College, London; Prof Camille Carroll, Principal Investigator — Newcastle University
Locations (2):
- United Kingdom (2):
  - UCLH, London
  - Clinical Ageing Research Unit, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing: Available on request Research teams may approach the MRC CTU with a formal data-sharing request detailing the specific requirement, proposed research, qualification of researchers and publication plan if they are interested in using EJS ACT-PD data. The request will be reviewed by the trial committees. Data and/or samples will be available for sharing following the end of a trial arm and the unblinding of participants. Researchers wishing to access the EJS ACT-PD Trial data should contact the Trial Management Group in the first instance. Following trial completion, requests for data and/ or sample sharing will be reviewed by an EJS ACT-PD access committee which will include the trial's Chief Investigators.

REFERENCES:
- See also: EJS ACT-PD Website — https://ejsactpd.com/